CLINICAL TRIAL: NCT06904833
Title: Assessment of Energy Expenditure of Elite Amateur Golfers Using a Buggy or Walking Over 2 Rounds of 18 Holes Using an ActiHeart® Monitor
Brief Title: Gauging Outcomes of Locomotion Formats
Acronym: GOLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24/SPS/075
Record Dates: First submitted 2025-03-17; First posted 2025-04-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Locomotor Activity
Keywords: energy expenditure; golf; actiheart; golf cart; performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walking (Active Comparator)
  Interventions: Device: locomotion formats
- Buggy (Active Comparator)
  Interventions: Device: locomotion formats

INTERVENTIONS:
Device: locomotion formats — two different types of popular locomotion methods in golf (i.e., walking 18 holes and using a buggy)

SUMMARY:
Investigators intend to use Actiheart® Monitors with a cohort of 16-30 elite amateur golfers over 18 (male and female) from Tournament Golf to clarify golfer's energy expenditure across a round of 18 holes in each condition at a championship course in Portugal.

In a randomised repeated measures design, participants will either walk or use a buggy for 18 holes. All sets of clubs will be placed in the buggy at all times. Baseline measures (e.g., weight, height, performance metrics, age will also be recorded). Each group will be assigned a helper/ coach to ensure only the correct participants are using the buggies. The buggy will be driven by a member of staff to ensure the buggy is moving at a controlled speed and only travelling to the necessary places on the golf course. Rounds will be timed from start to finish. Elements will be controlled throughout the week by the nutritionist on site. This includes practice sessions (e.g., driving range, chipping), gym sessions and the competitors will be playing under tournament conditions. Global positioning system (GPS) and step count will also be monitored.

Rate of perceived exertion (RPE) will also be measured using the modified Borg Scale . This will be collected pre round, during every 6 holes (holes 6, 12 and 18) and post round. Trackman (Trackman 4) machinery will also be set up every 6 holes (6, 12, 18), to measure performance variables (e.g., driving distance/ accuracy) at various points during the round to determine if there is a possible difference in performance when using a different method of transport. Players will not be told what these devices are measuring to ensure it doesn't affect mindset. Upgame will also be used to measure performance statistics and individuals scoring to determine if there is any correlation between this and energy expended. Force plates (Smart2move 1D) will also be used to measure ground reaction forces pre and post round by a strength and conditioning coach.

The principal investigator will transport the Actiheart ® monitors to Portugal. Prior to each round of 18 holes, participants will be fitted with an Actiheart® accelerometer (Actiheart®; dimensions: 39.7 × 30.3 ×9.25 mm; weight: 10.5 g) and chest heart rate monitor (Camn tech, Fenstanton, UK). Participant HR and activity levels will be recorded using 15 second epochs to estimate AEE for the duration of each activity and round of competitive golf. The data will be downloaded from the device immediately following each round and activity for analysis. The lead investigator will collect the data and then it will be analysed to establish the activity energy expenditure during a round of golf when walking or using a buggy.

Cognitive function measurements will also be assessed by a simplified version of VAS- Fatigue. We will use two visual rating scales (none to worst imaginable) pre and post round to measure cognitive fatigue and physical fatigue. A Stroop test will also be used to assess selective attention, inhibition and cognitive flexibility pre and post round. Players post round will be asked a 10-15 open ended questionnaire to assess their feelings towards using a buggy. Questions will include, 'did you think using the buggy today enhanced your performance?' and vice versa. The NASA- TLX. This measures mental demand, physical demand, temporal demand, performance, effort and frustration.

Differential RPE (d-RPE) will be asked of players post 18 holes which will allow us to quantify a perceived load for different subscales such as breathing, limb, cognitive/ technical and overall. Core temperature will be assessed using telemetry pills. Participants will swallow the pill at least one hour before we start getting a measure to ensure it has been digested. A reader will be used post round and held next to the participants stomach that will download all the relevant information. Data will be collected every 10 minutes for 60 minutes. To maximise the study's internal validity, all participants will be amateur golfers currently registered as students as the Tournament Golf College. The data will be collected and stored onto a secure LJMU drive, this will be pseudo- anonymised.

It is hoped that the result of this study will clarify energy expenditure of elite amateur male and female golfers whilst using a buggy or walking throughout a tournament week. This will allow players of all standards to implement practical nutrition strategies for fuelling and recovery and will confirm whether using a buggy may have positive implications for performance and health.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Elite Amateurs
* 18-50 years of age
* Handicaps 5 and below
* Members of Tournament Golf College (TGC)
* Physically active
* Healthy
* Injury Free
* Body weight >36.5kg

Exclusion Criteria:

* Gender/ Sex: Other
* Age: <18->50
* Injured/ Not competing
* Handicap >5
* Body weight <36.5kg
* Obstructive gastro-disease
* History of gastrointestinal surgery
* Current use of an implanted medical device
* Scheduled for an MRI scan during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure | during day 1 and day 2 of the 18 holes of golf.
  Measurement of activity energy expenditure using actiheart monitors using a buggy and walking

SECONDARY OUTCOMES:
Assessment of muscle force using force platforms | Day 1 and day 2 will include 18 holes of golf (one round). Testing will be done before and after these rounds.
Rate of perceived exertion | Day 1 and day 2 will include 18 holes of golf (one round). Testing will be done before and after these rounds and after every 6 holes.
driver swing speed using trackman | Day 1 and day 2 will include 18 holes of golf (one round). Testing will be done on the first hole of each round and every 6 holes.
Stroop colour word test | Day 1 and day 2 will include 18 holes of golf (one round). Testing will be done before and after these rounds.
NASA-TLX | Day 1 and day 2 will include 18 holes of golf (one round). Testing will be done after these rounds.
  The NASA Task Load Index scale will measure cognitive metrics (performance, temporal demand, mental demand, effort, frustration, physical demand). These are based on a scale of 1 (very low) to 20 (very high). The higher the score, the more challenging they found the round.
Core temperature using telemetry pills | Day 1 and day 2 will include 18 holes of golf (one round). Testing will be done before and after these rounds and after every 6 holes in these rounds.

CONTACTS AND LOCATIONS:
Locations (1):
- Tournament Golf College, Alcantarilha, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893